CLINICAL TRIAL: NCT05049577
Title: Can Preanesthetic Analgesia/Nociception Index (ANI) Predict Propofol Injection Pain
Brief Title: Preanesthetic Analgesia/Nociception Index (ANI) and Propofol Injection Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Cheol Lee,MD,PhD,, Professor, Wonkwang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: WonkwangUH8
Record Dates: First submitted 2021-08-24; First posted 2021-09-20 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Pain, Acute; Analgesia; Nociceptive Pain
MeSH Terms: conditions — Acute Pain; Agnosia; Nociceptive Pain | interventions — Analgesia

STUDY DESIGN:
Intervention Model Description: Prospective randomized and controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All study drugs were administered using a Minto pharmacokinetic model in a TCI device (Orchestra, Fresenius-Vial, France). The infusion pump was covered to blind the patients, investigator, and outcomes assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): To maintain blinding, in the control group, the remifentanil infusion was replaced with 50 ml of normal saline in 50 ml syringe. The remifentanil (or saline) infusion was run until the pump indicated the target Ce had been achieved. Pharmacokinetic model for remifentanil was the Minto model (Height, Weight, and Age) Anesthesia in all patients was induced using 2 mg/kg of 2% propofol. The attending anesthesiologist asked the patients how they felt pain to evaluate pain severity of PIP while half -dose of propofol was administered. After the rest of the propofol was administered, the attending anesthesiologists asked the same question.
  Interventions: Device: Analgesia/Nociception Index (ANI)
- Remifentanil group (Experimental): Remifentanil 1 mg was diluted into 50 ml of normal saline. A commercial TCI pump (Orchestra Base Primea, Fresenius Vial, France) was used for the effect-site TCI of remifentanil. The study groups received remifentanil to a target Ce of 4 ng/ ml. Pharmacokinetic model for remifentanil was the Minto model (Height, Weight, and Age) Anesthesia induction and the evaluation of pain were same as control group
  Interventions: Device: Analgesia/Nociception Index (ANI)

INTERVENTIONS:
Device: Analgesia/Nociception Index (ANI) — V1 and V5 electrocardiographic positions as per the manufacturer's recommendations. The ANI was continuously recorded and displayed with a frequency of 1 Hz. ANI scores measured immediately before propofol administration, half-dose administration (1mg/kg), and full-dose administration (2mg/kg)of propofol.
  Other Names: ANI MOC-9

SUMMARY:
Recently, Analgesia Nociception Index (ANI) has been evaluated for objectively measuring peri-operative pain and to guide intra-operative opioid administration during various surgeries.

Propofol injection pain (PIP) is a common problem and can be very distressing to the patient.

DETAILED DESCRIPTION:
This study aimed to the association of preanesthetic ANI scores and PIP in patients who scheduled for general anesthesia.

Before propofol administration in remifentanil group, preanesthetic ANI values (instant and mean) were checked after remifentanil to a target Ce of 4 ng/ml.

Control group received the same volume of saline as remifentanil group. Heart rate and bispectral index were checked as ANI. Point biserial correlation and ROC curve were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Male patients who scheduled for general anesthesia
* Cognitive patients who could understand this study

Exclusion Criteria:

* Patients receiving β-receptor blockers, ketamine, clonidine, or any vasoactive substance (i.e. metaraminol, ephedrine) and patients receiving neostigmine, atropine or glycopyrrolate.

Ages: 19 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male patients aged 19-60 years and the american society of anesthesiologists(ASA) class I or II who were scheduled for general anesthesia
Enrollment: 124 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The correlation of Analgesia/nociception Index (ANI) and Propofol injection pain (PIP) | Immediately before administration of propofol (2mg/kg)
  The correlation of preanesthetic ANI scores and incidence of PIP.

SECONDARY OUTCOMES:
Incidence and severity of PIP | during anesthesia induction ( half-dose (1mg/kg) and full-dose of (2mg/kg) propofol administration)
  Incidence and severity with numeric rating scales( 0= no pain, 100=worst pain) of propofol injection pain
The correlation of Analgesia/nociception Index (ANI) and Propofol injection pain (PIP) | Immediately before administration of propofol (2mg/kg)
  The correlation of preanesthetic ANI scores and severity of PIP.

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Lee, M.D,Ph.D, Principal Investigator — Department of anesthesiology and pain medicine
Locations (1):
- WonwangUH, Iksan, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No
if other researchers ask, a decision will be made after discussion with the co-authors

REFERENCES:
- [Background] Chanques G, Tarri T, Ride A, Prades A, De Jong A, Carr J, Molinari N, Jaber S. Analgesia nociception index for the assessment of pain in critically ill patients: a diagnostic accuracy study. Br J Anaesth. 2017 Oct 1;119(4):812-820. doi: 10.1093/bja/aex210. PMID 29121287
- [Background] Ledowski T. Objective monitoring of nociception: a review of current commercial solutions. Br J Anaesth. 2019 Aug;123(2):e312-e321. doi: 10.1016/j.bja.2019.03.024. Epub 2019 Apr 30. PMID 31047645
- [Background] Abdullayev R, Yildirim E, Celik B, Topcu Sarica L. Analgesia Nociception Index: Heart Rate Variability Analysis of Emotional Status. Cureus. 2019 Apr 2;11(4):e4365. doi: 10.7759/cureus.4365. PMID 31192070